CLINICAL TRIAL: NCT00093158
Title: The ACUITY Trial: A Randomized Comparison of Angiomax (Bivalirudin) Versus Heparin (Unfractionated Heparin or Enoxaparin) in Patients Undergoing Early Invasive Management for Acute Coronary Syndromes Without ST-Segment Elevation
Brief Title: Comparison of Angiomax Versus Heparin in Acute Coronary Syndromes (ACS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-02-08; ACUITY
Record Dates: First submitted 2004-10-04; First posted 2004-10-07 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Unstable Angina; Myocardial Infarction; Acute Disease
Keywords: Acute Coronary Syndromes
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction; Acute Disease; Acute Coronary Syndrome | interventions — bivalirudin; Anticoagulants

INTERVENTIONS:
Drug: Angiomax (bivalirudin) anticoagulant

SUMMARY:
The purpose of this study is to show that, when compared with heparin (enoxaparin or unfractionated heparin) and routine GPIIb/IIIa inhibition (either started upfront or at the time of percutaneous coronary intervention [PCI]; Arm A):

1. Bivalirudin with routine GPIIb/IIIa inhibition (either started upfront or at the time of PCI; Arm B) provides non-inferior or superior overall clinical outcomes and
2. Bivalirudin alone (Arm C) reduces clinically significant bleeding. An important secondary objective for this comparison is to show that bivalirudin is not inferior for ischemic complications.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged >=18 years at the time of randomization.
2. Have symptoms which include at least 10 minutes of angina or anginal equivalent that the investigator believes has a high likelihood of being ischemic in origin within the 24 hours prior to randomization consistent with a diagnosis of Unstable Angina/Non-ST Elevation Myocardial Infarction (UA/NSTEMI) (patients with symptoms atypical for cardiac ischemia should not be enrolled).
3. Meet at least one of the following criteria for UA/NSTEMI:

   1. All of the following four features: *Age >= to 65 years; *aspirin taken within the last 7 days; *two or more episodes of angina in the last 24 hours; *three or more of the following risk factors: hypertension, high cholesterol, family history, diabetes, current smoker OR
   2. ECG changes: New or presumably new ST-segment depression >=0.1 MV (>=1mm), or transient (<30 minutes) ST-segment elevation >=0.1MV (>=1mm) in at least 2 contiguous leads, OR
   3. Abnormal cardiac enzymes within the 24 hours before enrollment defined as elevated troponin I, T or creatine phosphokinase-MB isoenzyme (CPK-MB) level greater than the site's upper limit of normal (ULN) OR
   4. History of coronary artery disease with documentation of one of the following: *prior angiography (coronary stenosis of >50%); *prior PCI or Coronary Artery Bypass Grafting (CABG); *prior definite, documented myocardial infarction.
4. Provide written informed consent before initiation of any study related procedures.

Exclusion Criteria:

1. Anticipated inability to perform angiography within 72 hours of randomization and anticipated inability to perform any intervention required (PCI or CABG) within the index hospitalization.
2. ST segment elevation of >1 mm in 2 contiguous ECG leads lasting for >30 minutes, or new left bundle branch block, or a clinical syndrome consistent with acute evolving transmural MI requiring immediate thrombolytic or interventional reperfusion therapy.
3. Cardiogenic shock (systolic blood pressure <80 mmHg for >30 minutes not responding to intravenous fluids, or requiring intravenous pressor agents or an intra-aortic balloon pump).
4. Bleeding diathesis or any history of hemorrhagic stroke or other intra-cerebral bleed, cerebral arteriovenous malformation, cerebral aneurysm or prior ischemic stroke within the last 2 years, or any prior stroke with residual neurologic deficit. Gastrointestinal or genitourinary bleeding within the last 2-weeks.
5. Platelet count <100,000 cells/mm3 at baseline, or history of heparin induced thrombocytopenia
6. Patients on warfarin or phenprocoumon, unless they can be safely discontinued and the baseline INR is < 1.5 times control.
7. Allergy to pork or pork products.
8. Patients who have been started on and received 2 or more doses of low molecular weight heparin for the current admission prior to randomization (patients who have received one dose of low molecular weight heparin may still be enrolled.
9. Patients who have been started on bivalirudin in the 6 hours prior to randomization
10. Thrombolytic therapy or abciximab use within the last 24 hours.
11. Treatment with a GPIIb/IIIa inhibitor at the time of randomization, which cannot be discontinued.
12. Patients on Arixtra (fondaparinux).
13. Absolute contraindication or allergy to:

    * any one of enoxaparin, unfractionated heparin, bivalirudin or aspirin
    * both abciximab and eptifibatide
    * both eptifibatide and tirofiban
    * iodinated contrast which cannot be pre-medicated
14. Contraindications to angiography, including but not limited to severe peripheral vascular disease.
15. Angina from secondary causes.
16. Pregnancy or nursing mothers. Women of child bearing potential must have a negative urine or serum pregnancy test prior to enrollment.
17. Calculated serum creatinine clearance < 30 mL/min (Determined by the Cockcroft Gault formula: ((140-age in yrs) x weight in kg)/(814.464 x Creatinine in mmol/l) or /(72 x [Creatinine in mg/dL]). For women, multiply by 0.85.
18. Previous enrollment in this study.
19. Patients currently enrolled in another investigational drug study that has not completed the follow-up phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13800
Dates: Start 2003-08; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Research Foundation, New York, New York, United States

REFERENCES:
- [Derived] Redfors B, Kirtane AJ, Pocock SJ, Ayele GM, Deliargyris EN, Mehran R, Stone GW, Genereux P. Bleeding Events Before Coronary Angiography in Patients With Non-ST-Segment Elevation Acute Coronary Syndrome. J Am Coll Cardiol. 2016 Dec 20;68(24):2608-2618. doi: 10.1016/j.jacc.2016.09.957. PMID 27978944
- [Derived] Giacoppo D, Madhavan MV, Baber U, Warren J, Bansilal S, Witzenbichler B, Dangas GD, Kirtane AJ, Xu K, Kornowski R, Brener SJ, Genereux P, Stone GW, Mehran R. Impact of Contrast-Induced Acute Kidney Injury After Percutaneous Coronary Intervention on Short- and Long-Term Outcomes: Pooled Analysis From the HORIZONS-AMI and ACUITY Trials. Circ Cardiovasc Interv. 2015 Aug;8(8):e002475. doi: 10.1161/CIRCINTERVENTIONS.114.002475. PMID 26198286
- [Derived] Ben-Gal Y, Mohr R, Feit F, Ohman EM, Kirtane A, Xu K, Mehran R, Stone GW. Surgical versus percutaneous coronary revascularization for multivessel disease in diabetic patients with non-ST-segment-elevation acute coronary syndrome: analysis from the Acute Catheterization and Early Intervention Triage Strategy trial. Circ Cardiovasc Interv. 2015 Jun;8(6):e002032. doi: 10.1161/CIRCINTERVENTIONS.114.002032. PMID 26019142
- [Derived] Genereux P, Bernard S, Palmerini T, Caixeta A, Rosner G, Reiss GR, Xu K, Mehran R, Stone GW; ACUITY Trial Investigators. Incidence, predictors, and impact of neurological events in non-ST-segment elevation acute coronary syndromes: the ACUITY trial. EuroIntervention. 2015 Aug;11(4):399-406. doi: 10.4244/EIJY14M07_06. PMID 25022226
- [Derived] Planer D, Mehran R, Ohman EM, White HD, Newman JD, Xu K, Stone GW. Prognosis of patients with non-ST-segment-elevation myocardial infarction and nonobstructive coronary artery disease: propensity-matched analysis from the Acute Catheterization and Urgent Intervention Triage Strategy trial. Circ Cardiovasc Interv. 2014 Jun;7(3):285-93. doi: 10.1161/CIRCINTERVENTIONS.113.000606. Epub 2014 May 20. PMID 24847016
- [Derived] Robertson JO, Ebrahimi R, Lansky AJ, Mehran R, Stone GW, Lincoff AM. Impact of cigarette smoking on extent of coronary artery disease and prognosis of patients with non-ST-segment elevation acute coronary syndromes: an analysis from the ACUITY Trial (Acute Catheterization and Urgent Intervention Triage Strategy). JACC Cardiovasc Interv. 2014 Apr;7(4):372-9. doi: 10.1016/j.jcin.2013.11.017. Epub 2014 Mar 14. PMID 24630881
- [Derived] Genereux P, Madhavan MV, Mintz GS, Maehara A, Palmerini T, Lasalle L, Xu K, McAndrew T, Kirtane A, Lansky AJ, Brener SJ, Mehran R, Stone GW. Ischemic outcomes after coronary intervention of calcified vessels in acute coronary syndromes. Pooled analysis from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) and ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) TRIALS. J Am Coll Cardiol. 2014 May 13;63(18):1845-54. doi: 10.1016/j.jacc.2014.01.034. Epub 2014 Feb 19. PMID 24561145
- [Derived] Madhavan MV, Genereux P, Rubin J, Palmerini T, Caixeta A, Xu K, Weisz G, Mehran R, Stone GW. Usefulness of the SYNTAX score to predict acute kidney injury after percutaneous coronary intervention (from the Acute Catheterization and Urgent Intervention Triage Strategy Trial). Am J Cardiol. 2014 Apr 15;113(8):1331-7. doi: 10.1016/j.amjcard.2013.12.041. Epub 2014 Jan 31. PMID 24560063
- [Derived] Meier P, Lansky AJ, Fahy M, Xu K, White HD, Bertrand ME, Mehran R, Stone GW. The impact of the coronary collateral circulation on outcomes in patients with acute coronary syndromes: results from the ACUITY trial. Heart. 2014 Apr;100(8):647-51. doi: 10.1136/heartjnl-2013-304435. Epub 2013 Dec 5. PMID 24310521
- [Derived] Ertelt K, Genereux P, Mintz GS, Reiss GR, Kirtane AJ, Madhavan MV, Fahy M, Williams MR, Brener SJ, Mehran R, Stone GW. Impact of the severity of coronary artery calcification on clinical events in patients undergoing coronary artery bypass grafting (from the Acute Catheterization and Urgent Intervention Triage Strategy Trial). Am J Cardiol. 2013 Dec 1;112(11):1730-7. doi: 10.1016/j.amjcard.2013.07.038. Epub 2013 Sep 5. PMID 24012035
- [Derived] Palmerini T, Genereux P, Caixeta A, Cristea E, Lansky A, Mehran R, Della Riva D, Fahy M, Xu K, Stone GW. A new score for risk stratification of patients with acute coronary syndromes undergoing percutaneous coronary intervention: the ACUITY-PCI (Acute Catheterization and Urgent Intervention Triage Strategy-Percutaneous Coronary Intervention) risk score. JACC Cardiovasc Interv. 2012 Nov;5(11):1108-16. doi: 10.1016/j.jcin.2012.07.011. PMID 23174634
- [Derived] Dangas GD, Claessen BE, Mehran R, Xu K, Fahy M, Parise H, Henriques JP, Ohman EM, White HD, Stone GW. Development and validation of a stent thrombosis risk score in patients with acute coronary syndromes. JACC Cardiovasc Interv. 2012 Nov;5(11):1097-105. doi: 10.1016/j.jcin.2012.07.012. PMID 23174632
- [Derived] Ndrepepa G, Neumann FJ, Deliargyris EN, Mehran R, Mehilli J, Ferenc M, Schulz S, Schomig A, Kastrati A, Stone GW. Bivalirudin versus heparin plus a glycoprotein IIb/IIIa inhibitor in patients with non-ST-segment elevation myocardial infarction undergoing percutaneous coronary intervention after clopidogrel pretreatment: pooled analysis from the ACUITY and ISAR-REACT 4 trials. Circ Cardiovasc Interv. 2012 Oct;5(5):705-12. doi: 10.1161/CIRCINTERVENTIONS.112.972869. Epub 2012 Oct 9. PMID 23048052
- [Derived] Rosner GF, Kirtane AJ, Genereux P, Lansky AJ, Cristea E, Gersh BJ, Weisz G, Parise H, Fahy M, Mehran R, Stone GW. Impact of the presence and extent of incomplete angiographic revascularization after percutaneous coronary intervention in acute coronary syndromes: the Acute Catheterization and Urgent Intervention Triage Strategy (ACUITY) trial. Circulation. 2012 May 29;125(21):2613-20. doi: 10.1161/CIRCULATIONAHA.111.069237. Epub 2012 May 1. PMID 22550156
- [Derived] Genereux P, Palmerini T, Caixeta A, Rosner G, Green P, Dressler O, Xu K, Parise H, Mehran R, Serruys PW, Stone GW. Quantification and impact of untreated coronary artery disease after percutaneous coronary intervention: the residual SYNTAX (Synergy Between PCI with Taxus and Cardiac Surgery) score. J Am Coll Cardiol. 2012 Jun 12;59(24):2165-74. doi: 10.1016/j.jacc.2012.03.010. Epub 2012 Apr 4. PMID 22483327
- [Derived] Stone GW, Clayton TC, Mehran R, Dangas G, Parise H, Fahy M, Pocock SJ. Impact of major bleeding and blood transfusions after cardiac surgery: analysis from the Acute Catheterization and Urgent Intervention Triage strategY (ACUITY) trial. Am Heart J. 2012 Mar;163(3):522-9. doi: 10.1016/j.ahj.2011.11.016. PMID 22424026
- [Derived] Acharji S, Baber U, Mehran R, Fahy M, Kirtane AJ, Lansky AJ, Stone GW. Prognostic significance of elevated baseline troponin in patients with acute coronary syndromes and chronic kidney disease treated with different antithrombotic regimens: a substudy from the ACUITY trial. Circ Cardiovasc Interv. 2012 Apr;5(2):157-65. doi: 10.1161/CIRCINTERVENTIONS.111.963876. Epub 2012 Feb 21. PMID 22354934
- [Derived] Palmerini T, Dangas G, Mehran R, Caixeta A, Genereux P, Fahy MP, Xu K, Cristea E, Lansky AJ, Stone GW. Predictors and implications of stent thrombosis in non-ST-segment elevation acute coronary syndromes: the ACUITY Trial. Circ Cardiovasc Interv. 2011 Dec 1;4(6):577-84. doi: 10.1161/CIRCINTERVENTIONS.111.963884. Epub 2011 Oct 25. PMID 22028471
- [Derived] Palmerini T, Genereux P, Caixeta A, Cristea E, Lansky A, Mehran R, Dangas G, Lazar D, Sanchez R, Fahy M, Xu K, Stone GW. Prognostic value of the SYNTAX score in patients with acute coronary syndromes undergoing percutaneous coronary intervention: analysis from the ACUITY (Acute Catheterization and Urgent Intervention Triage StrategY) trial. J Am Coll Cardiol. 2011 Jun 14;57(24):2389-97. doi: 10.1016/j.jacc.2011.02.032. PMID 21658558
- [Derived] Caixeta A, Dangas GD, Mehran R, Feit F, Nikolsky E, Lansky AJ, Aoki J, Moses JW, Steinhubl SR, White HD, Ohman EM, Manoukian SV, Fahy M, Stone GW. Incidence and clinical consequences of acquired thrombocytopenia after antithrombotic therapies in patients with acute coronary syndromes: results from the Acute Catheterization and Urgent Intervention Triage Strategy (ACUITY) trial. Am Heart J. 2011 Feb;161(2):298-306.e1. doi: 10.1016/j.ahj.2010.10.035. PMID 21315212
- [Derived] Ben-Gal Y, Moses JW, Mehran R, Lansky AJ, Weisz G, Nikolsky E, Argenziano M, Williams MR, Colombo A, Aylward PE, Stone GW. Surgical versus percutaneous revascularization for multivessel disease in patients with acute coronary syndromes: analysis from the ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) trial. JACC Cardiovasc Interv. 2010 Oct;3(10):1059-67. doi: 10.1016/j.jcin.2010.06.017. PMID 20965465
- [Derived] Caixeta A, Stone GW, Mehran R, Lee EA, McLaurin BT, Cox DA, Bertrand ME, Lincoff AM, Moses JW, White HD, Ohman EM, Palmerini T, Syros G, Kittas C, Fahy M, Hooper WC, Lansky AJ, Dangas GD. Predictive value of C-reactive protein on 30-day and 1-year mortality in acute coronary syndromes: an analysis from the ACUITY trial. J Thromb Thrombolysis. 2011 Feb;31(2):154-64. doi: 10.1007/s11239-010-0516-y. PMID 20953817
- [Derived] Lansky AJ, Goto K, Cristea E, Fahy M, Parise H, Feit F, Ohman EM, White HD, Alexander KP, Bertrand ME, Desmet W, Hamon M, Mehran R, Moses J, Leon M, Stone GW. Clinical and angiographic predictors of short- and long-term ischemic events in acute coronary syndromes: results from the Acute Catheterization and Urgent Intervention Triage strategY (ACUITY) trial. Circ Cardiovasc Interv. 2010 Aug;3(4):308-16. doi: 10.1161/CIRCINTERVENTIONS.109.887604. Epub 2010 Jul 20. PMID 20647564
- [Derived] Goto K, Lansky AJ, Fahy M, Cristea E, Feit F, Ohman EM, White HD, Alexander KP, Bertrand ME, Desmet W, Hamon M, Mehran R, Stone GW. Predictors of outcomes in medically treated patients with acute coronary syndromes after angiographic triage: an Acute Catheterization And Urgent Intervention Triage Strategy (ACUITY) substudy. Circulation. 2010 Feb 23;121(7):853-62. doi: 10.1161/CIRCULATIONAHA.109.877944. Epub 2010 Feb 8. PMID 20142447
- [Derived] Sanborn TA, Ebrahimi R, Manoukian SV, McLaurin BT, Cox DA, Feit F, Hamon M, Mehran R, Stone GW. Impact of femoral vascular closure devices and antithrombotic therapy on access site bleeding in acute coronary syndromes: The Acute Catheterization and Urgent Intervention Triage Strategy (ACUITY) trial. Circ Cardiovasc Interv. 2010 Feb 1;3(1):57-62. doi: 10.1161/CIRCINTERVENTIONS.109.896704. Epub 2010 Jan 26. PMID 20118151
- [Derived] Pocock SJ, Mehran R, Clayton TC, Nikolsky E, Parise H, Fahy M, Lansky AJ, Bertrand ME, Lincoff AM, Moses JW, Ohman EM, White HD, Stone GW. Prognostic modeling of individual patient risk and mortality impact of ischemic and hemorrhagic complications: assessment from the Acute Catheterization and Urgent Intervention Triage Strategy trial. Circulation. 2010 Jan 5;121(1):43-51. doi: 10.1161/CIRCULATIONAHA.109.878017. Epub 2009 Dec 21. PMID 20026777
- [Derived] Prasad A, Gersh BJ, Bertrand ME, Lincoff AM, Moses JW, Ohman EM, White HD, Pocock SJ, McLaurin BT, Cox DA, Lansky AJ, Mehran R, Stone GW. Prognostic significance of periprocedural versus spontaneously occurring myocardial infarction after percutaneous coronary intervention in patients with acute coronary syndromes: an analysis from the ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) trial. J Am Coll Cardiol. 2009 Jul 28;54(5):477-86. doi: 10.1016/j.jacc.2009.03.063. PMID 19628125
- [Derived] Lincoff AM, Steinhubl SR, Manoukian SV, Chew D, Pollack CV Jr, Feit F, Ware JH, Bertrand ME, Ohman EM, Desmet W, Cox DA, Mehran R, Stone GW; Acute Catheterization and Urgent Intervention Triage strategY of Trial Investigators. Influence of timing of clopidogrel treatment on the efficacy and safety of bivalirudin in patients with non-ST-segment elevation acute coronary syndromes undergoing percutaneous coronary intervention: an analysis of the ACUITY (Acute Catheterization and Urgent Intervention Triage strategY) trial. JACC Cardiovasc Interv. 2008 Dec;1(6):639-48. doi: 10.1016/j.jcin.2008.10.004. PMID 19463378
- [Derived] Ebrahimi R, Dyke C, Mehran R, Manoukian SV, Feit F, Cox DA, Gersh BJ, Ohman EM, White HD, Moses JW, Ware JH, Lincoff AM, Stone GW. Outcomes following pre-operative clopidogrel administration in patients with acute coronary syndromes undergoing coronary artery bypass surgery: the ACUITY (Acute Catheterization and Urgent Intervention Triage strategY) trial. J Am Coll Cardiol. 2009 May 26;53(21):1965-72. doi: 10.1016/j.jacc.2009.03.006. PMID 19460609
- [Derived] Lopes RD, Alexander KP, Manoukian SV, Bertrand ME, Feit F, White HD, Pollack CV Jr, Hoekstra J, Gersh BJ, Stone GW, Ohman EM. Advanced age, antithrombotic strategy, and bleeding in non-ST-segment elevation acute coronary syndromes: results from the ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) trial. J Am Coll Cardiol. 2009 Mar 24;53(12):1021-30. doi: 10.1016/j.jacc.2008.12.021. PMID 19298914
- [Derived] Aoki J, Lansky AJ, Mehran R, Moses J, Bertrand ME, McLaurin BT, Cox DA, Lincoff AM, Ohman EM, White HD, Parise H, Leon MB, Stone GW. Early stent thrombosis in patients with acute coronary syndromes treated with drug-eluting and bare metal stents: the Acute Catheterization and Urgent Intervention Triage Strategy trial. Circulation. 2009 Feb 10;119(5):687-98. doi: 10.1161/CIRCULATIONAHA.108.804203. Epub 2009 Jan 26. PMID 19171852
- [Derived] Pinto DS, Stone GW, Shi C, Dunn ES, Reynolds MR, York M, Walczak J, Berezin RH, Mehran R, McLaurin BT, Cox DA, Ohman EM, Lincoff AM, Cohen DJ; ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) Investigators. Economic evaluation of bivalirudin with or without glycoprotein IIb/IIIa inhibition versus heparin with routine glycoprotein IIb/IIIa inhibition for early invasive management of acute coronary syndromes. J Am Coll Cardiol. 2008 Nov 25;52(22):1758-68. doi: 10.1016/j.jacc.2008.08.021. PMID 19022155
- [Derived] Stone GW, Ware JH, Bertrand ME, Lincoff AM, Moses JW, Ohman EM, White HD, Feit F, Colombo A, McLaurin BT, Cox DA, Manoukian SV, Fahy M, Clayton TC, Mehran R, Pocock SJ; ACUITY Investigators. Antithrombotic strategies in patients with acute coronary syndromes undergoing early invasive management: one-year results from the ACUITY trial. JAMA. 2007 Dec 5;298(21):2497-506. doi: 10.1001/jama.298.21.2497. PMID 18056903
- [Derived] Stone GW, White HD, Ohman EM, Bertrand ME, Lincoff AM, McLaurin BT, Cox DA, Pocock SJ, Ware JH, Feit F, Colombo A, Manoukian SV, Lansky AJ, Mehran R, Moses JW; Acute Catheterization and Urgent Intervention Triage strategy (ACUITY) trial investigators. Bivalirudin in patients with acute coronary syndromes undergoing percutaneous coronary intervention: a subgroup analysis from the Acute Catheterization and Urgent Intervention Triage strategy (ACUITY) trial. Lancet. 2007 Mar 17;369(9565):907-19. doi: 10.1016/S0140-6736(07)60450-4. PMID 17368152
- [Derived] Stone GW, Bertrand ME, Moses JW, Ohman EM, Lincoff AM, Ware JH, Pocock SJ, McLaurin BT, Cox DA, Jafar MZ, Chandna H, Hartmann F, Leisch F, Strasser RH, Desaga M, Stuckey TD, Zelman RB, Lieber IH, Cohen DJ, Mehran R, White HD; ACUITY Investigators. Routine upstream initiation vs deferred selective use of glycoprotein IIb/IIIa inhibitors in acute coronary syndromes: the ACUITY Timing trial. JAMA. 2007 Feb 14;297(6):591-602. doi: 10.1001/jama.297.6.591. PMID 17299194
- [Derived] Stone GW, McLaurin BT, Cox DA, Bertrand ME, Lincoff AM, Moses JW, White HD, Pocock SJ, Ware JH, Feit F, Colombo A, Aylward PE, Cequier AR, Darius H, Desmet W, Ebrahimi R, Hamon M, Rasmussen LH, Rupprecht HJ, Hoekstra J, Mehran R, Ohman EM; ACUITY Investigators. Bivalirudin for patients with acute coronary syndromes. N Engl J Med. 2006 Nov 23;355(21):2203-16. doi: 10.1056/NEJMoa062437. PMID 17124018